CLINICAL TRIAL: NCT02876393
Title: A Systematic Study of Retinal Structure and Function in Diabetic Macular Oedema
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Usha Chakravarthy, Professor, Queen's University, Belfast
Other Study IDs: 14/NI/1025
Record Dates: First submitted 2016-04-28; First posted 2016-08-23 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Persons with type 1 or type 2 DM with features of DR and or DMO ranging from extremely mild to severe.
- Control definition: Persons with a history of type 1 or type 2 DM without any clinical features of DR or DMO in either eye or persons without a history of DM and without retinal disease in either eye.

SUMMARY:
Diabetic retinopathy(DR) is a sight threatening condition that occurs in persons with diabetes. DR arises as a consequence of damage to the retinal blood vessels and is related to the high and fluctuating sugar levels in the blood stream. An eye with DR will have abnormal appearing retinal blood vessels which become engorged and dilated, leaky and fragile or undergo closure. The net result is a picture of haemorrhage and or ischaemia (lack of blood supply). A particular feature of DR is the accumulation of fluid in the macula which is the central part of the retina and responsible for detailed eye sight. This peculiar form of DR is called Diabetic Macular Oedema (DMO). DMO can occur in isolation without other features of DR. DMO is commoner in type 2 diabetes where insulin resistance and abnormalities of blood fats are found. The investigators wish to study DR and DMO using high resolution retinal imaging and functional tests in normal participants, those participants with diabetes without any overt signs of disease and those with DR and DMO in order to understand how the condition develops and whether there are any unique risk factors that can be identified

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Healthy controls without DM):

* Persons older than 18 years without DM
* Fundus free of any signs of retinal disease
* Best Corrected Visual Acuity of 20/40 (73 ETDRS letters) in both eyes

Group 2 (Persons with DM with no retinopathy):

* Persons with Type 1 or type 2 diabetes older than 18 years
* Normal fundus, Absence of features of DR or DMO in both eyes
* Best Corrected Visual Acuity 20/40 (73 ETDRS letters) in at least one eye

Group 3:

* Persons with Type 1 or type 2 diabetes 18 years and older
* Fundus signs of mild, moderate or severe DR and or DMO
* Best Corrected Visual Acuity 20/200 (33 ETDRS letters) or better

Exclusion Criteria:

* Recent ocular surgical procedures performed within the previous 3 months
* Presence of ocular confounding disorders such as neovascular age related macular degeneration, glaucoma or active uveitis
* Serious life threatening conditions that would preclude attendance in the longitudinal part of the study
* Neurological conditions that can impair vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants with DR of different severity levels ranging from minimal DR to severe DR with or without DMO who attend the diabetic clinics will be invited to participate. Opportunistic sampling will be used to ensure that the different severity levels of DR and or DMO will be adequately represented.The Northern Ireland Cohort Longitudinal Study On ageing (NICOLA), a non-interventional epidemiological study of healthy ageing in older adults aged 50 years and above has commenced and is currently recruiting some 8500 participants. Participants in NICOLA who are known to have DM or have been recently diagnosed with DM will be approached and asked if willing to return for detailed functional testing of the eye. This will supplement the group with DM but with no changes of DR.
  Control participants with DM but without DR will be recruited from the metabolic clinics of the Belfast Trust.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Presence of DMO evaluated from the optical coherence tomography (OCT) images | The outcome measures will be assessed at the end of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Usha Chakravarthy, Phd FRCopth, Principal Investigator — Queens University Belfast
Locations (1):
- NI clinical Research Facility,51 Lisburn Road, Belfast, United Kingdom